CLINICAL TRIAL: NCT01273818
Title: Is Topical Antibiotic Prophylaxis Effective in Lichtenstein Hernia Repair: a Comparison Study
Brief Title: Effectiveness of Topical Antibiotic Prophylaxis in Inguinal Hernia Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Diskapi Teaching and Research Hospital (Other)
Responsible Party: Principal Investigator, Duray Seker, M.D. Surgery, Diskapi Teaching and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FC-001
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Results first posted 2014-12-29 (Estimated); Last update posted 2014-12-29 (Estimated); Status verified 2014-09

CONDITIONS: Inguinal Hernia
Keywords: inguinal hernia; infection prophylaxis; topical gentamicin
MeSH Terms: conditions — Hernia, Inguinal | interventions — Gentamicins; Cefazolin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- gentamicin (Active Comparator): 80 mg gentamicin topical application intraoperatively
  Interventions: Drug: Gentamicin
- Cefazolin (Active Comparator): Application of 1000 mg cefazolin intra venously 1 hour before surgery
  Interventions: Drug: Cefazolin
- gentamicin and cefazolin (Active Comparator): 1000 mg cefazolin application 1 hour before surgery and topical 80 mg gentamicin intraoperatively
  Interventions: Drug: Gentamicin and cefazolin

INTERVENTIONS:
Drug: Gentamicin and cefazolin — 80 mg topically, intra-operative,single dose and intravenous 1000 mg cefazolin 1 hour before operation
  Other Names: Drug: Cefazolin; Other names:; Cezol; Eqizolin; Drug: Gentamicin; Gensif; Gentamed
  Arms: gentamicin and cefazolin
Drug: Cefazolin — 1000 mg cefazolin application intravenously 1 hour before operation
  Other Names: Cezal; Eqizolin
  Arms: Cefazolin
Drug: Gentamicin — 80 mg gentamicin application intraoperatively
  Other Names: Gensif; Gentamed
  Arms: gentamicin

SUMMARY:
Aim of this study is to measure the effectiveness of topical gentamicin to prevent post-operative infection in inguinal tension-free hernia repair operation.Secondary aim is, if it is effective as a prophylactic agent, to compare it's effect with intra venous single dose cefazolin sodium prophylaxis.

DETAILED DESCRIPTION:
This study is a single blind prospective randomized trial. To measure and compare the effectiveness intra-operative topical gentamicin application in tension-free inguinal hernia repair in contrast to intravenous peri-operative prophylactic cefazolin sodium and combination of gentamicin and cephazolin this study is designed.

The patients are grouped randomly in to two groups:

* Group1;intravenous cefazolin sodium
* Group2;topical gentamicin
* Group3:topical gentamicin and intravenous cefazolin sodium

As a control group we decided to use the data of control groups ( without any prophylactic agent usage ) of previous studies done in our clinic and medical data base reviews.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of inguinal hernia

Exclusion Criteria:

* Femoral hernia
* Emergency cases

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2011-01; Primary Completion 2013-02 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gaye E Seker, MD, Principal Investigator — Diskapi Yildirim Beyazit Teaching and research Hospital; Duray Seker, MD, Study Director — Diskapi Yildirim Beyazit Teaching and research Hospital; Bahattin Bayar, MD, Study Chair — Diskapi Yildirim Beyazit Teaching and research Hospital; Zafer Ergul, MD, Study Chair — Diskapi Yildirim Beyazit Teaching and research Hospital; Hakan Kulacoglu, Professor, Study Chair — Diskapi Yildirim Beyazit Teaching and research Hospital
Locations (1):
- Diskapi Yildirim Beyazit Teaching and research Hospital, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Pessaux P, Lermite E, Blezel E, Msika S, Hay JM, Flamant Y, Deepak V, Arnaud JP; French Associations for Surgical Research. Predictive risk score for infection after inguinal hernia repair. Am J Surg. 2006 Aug;192(2):165-71. doi: 10.1016/j.amjsurg.2006.05.003. PMID 16860624
- [Background] Tzovaras G, Delikoukos S, Christodoulides G, Spyridakis M, Mantzos F, Tepetes K, Athanassiou E, Hatzitheofilou C. The role of antibiotic prophylaxis in elective tension-free mesh inguinal hernia repair: results of a single-centre prospective randomised trial. Int J Clin Pract. 2007 Feb;61(2):236-9. doi: 10.1111/j.1742-1241.2006.00977.x. PMID 16930145
- [Background] Zuvela M, Milicevic M, Galun D, Lekic N, Basaric D, Tomic D, Petrovic M, Palibrk I. [Infection in hernia surgery]. Acta Chir Iugosl. 2005;52(1):9-26. doi: 10.2298/aci0501009z. Serbian. PMID 16119310
- [Background] Praveen S, Rohaizak M. Local antibiotics are equivalent to intravenous antibiotics in the prevention of superficial wound infection in inguinal hernioplasty. Asian J Surg. 2009 Jan;32(1):59-63. doi: 10.1016/S1015-9584(09)60011-7. PMID 19321405
- [Background] Aufenacker TJ, Koelemay MJ, Gouma DJ, Simons MP. Systematic review and meta-analysis of the effectiveness of antibiotic prophylaxis in prevention of wound infection after mesh repair of abdominal wall hernia. Br J Surg. 2006 Jan;93(1):5-10. doi: 10.1002/bjs.5186. PMID 16252314
- [Background] Shankar VG, Srinivasan K, Sistla SC, Jagdish S. Prophylactic antibiotics in open mesh repair of inguinal hernia - a randomized controlled trial. Int J Surg. 2010;8(6):444-7. doi: 10.1016/j.ijsu.2010.05.011. Epub 2010 Jun 9. PMID 20538079
- [Background] Aufenacker TJ, van Geldere D, van Mesdag T, Bossers AN, Dekker B, Scheijde E, van Nieuwenhuizen R, Hiemstra E, Maduro JH, Juttmann JW, Hofstede D, van Der Linden CT, Gouma DJ, Simons MP. The role of antibiotic prophylaxis in prevention of wound infection after Lichtenstein open mesh repair of primary inguinal hernia: a multicenter double-blind randomized controlled trial. Ann Surg. 2004 Dec;240(6):955-60; discussion 960-1. doi: 10.1097/01.sla.0000145926.74300.42. PMID 15570201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period begins in Jan 2011. This period will be completed when record of minimum number participants ( according to power analysis) in each arm is completed.Location is surgery clinic of our hospital.
Pre-assignment Details: Totaly, 24 patients who were known using any kind of antibiotics for any reason just prior to surgery or just after the surgery and having history of allergic reactions to antibiotics used in this study were excluded.
Groups:
- Gentamicin: Gentamicin arm: application of 80 mg gentamycin topically
- Cefazolin: Application of 1000 mg cefazolin sodium intra venously 1 hour before surgery
- Gentamicin+ Cefazolin Sodium: Application of intravenous 1000 mg cefazolin sodium 1 hour before surgery + topical 80 mg gentamicin intraoperatively
Period: Overall Study
Arm/Group | Gentamicin | Cefazolin | Gentamicin+ Cefazolin Sodium
Started | 100 | 100 | 100
Completed | 87 | 98 | 91
Not Completed | 13 | 2 | 9
Not completed — Physician Decision | 13 | 2 | 9

BASELINE CHARACTERISTICS:
Population: 300 consequtive patients were diveded into three groups randomly, but during follow-up period since 24 patients used any kind of antibiotics for reasons other than postoperative complications, only 276 patients were analyzed.
Groups:
- Cephazolin: Application of 1000 mg cefazolin sodium intra venously 1 hour before surgery
- Total: Total of all reporting groups
Arm/Group | Gentamicin | Cephazolin | Gentamicin+ Cefazolin Sodium | Total
Number analyzed (Participants) | 87 | 98 | 91 | 276
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 60 | 65 | 71 | 196
  >=65 years | 27 | 33 | 20 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.39 (15.39) | 49.60 (13.85) | 50.36 (15.49) | 50.10 (14.85)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 5 | 5 | 17
  Male | 80 | 93 | 86 | 259
Region of Enrollment [Number; unit: participants]
  Turkey | 87 | 98 | 91 | 276

OUTCOME MEASURES:

1. Primary Outcome: Rate of Post-operative Infection
Time Frame: within the first 30 days after surgery
Reporting Status: Not Posted

2. Primary Outcome: Number of Infections in Each Study Arm
Description: Patients were examined on postoperative 30 days for the presence of surgical site infection.
Time Frame: within the 30 days after surgery
Measure: Number; unit: infections
Groups:
- Topical Gentamicin: Total number of patients to which topical gentamicin was applied for prophylaxis
- Cefazolin IV: Total number of patients to which ceephazoline (İV) was applied for prophylaxis
- Topical and iv: Total number of patients to which topical gentamicin and cephazoline (iv) was applied for prophylaxis
Arm/Group | Topical Gentamicin | Cefazolin IV | Topical and iv
Number analyzed (Participants) | 87 | 98 | 91
infections | 1 | 3 | 0
Statistical Analysis 1: Comparison: Topical Gentamicin vs Cefazolin IV; Comparison Group Selection: our primary outcome is "infection positive or negative"so, we compared the frequencies of being positive infections for these three groups. Our null hypothesis is " positive infection frequencies are same for three groups". We calculated post-hoc power for this design and found 0.99 for the percentages which shows positive infections respectively for Topical Gentamicin, cefazoline iv and topical gentamicin and iv cefazolin; 2.3%, 3.1% and 0%; Test type: Superiority or Other; p = 0.198, Fisher Exact; Fscher exact test — we did not need an estimation parameter such as odds or relative risk because of our experimental design and hypothesis of this study

ADVERSE EVENTS:
Groups:
- Gentamicin: Gentamicin arm: application of 80 mg gentamycin topically
  Gentamicins+cephazolin sodium: 80 mg topically, intra-operative,single dose
  No adverse effect
- Cephazolin: Application of 1000 mg cefazolin sodium intra venously 1 hour before surgery
  Gentamicins+cephazolin sodium: 80 mg topically, intra-operative,single dose
  No adverse effect
- Gentamicin+ Cefazolin Sodium: Application of intravenous 1000 mg cefazolin sodium 1 hour before surgery + topical 80 mg gentamicin intraoperatively
  Gentamicins+cephazolin sodium: 80 mg topically, intra-operative,single dose
  No adverse effect
Arm/Group | Gentamicin | Cephazolin | Gentamicin+ Cefazolin Sodium
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/98 | 0/91
Other Adverse Events (participants affected / at risk) | 0/87 | 0/98 | 0/91

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No